CLINICAL TRIAL: NCT00867529
Title: Addition of Pre- and Post-Transplant Rituximab for Patients Undergoing Non-myeloablative Allogeneic Hematopoietic Cell Transplantation With Relapsed or Refractory CD20+ B-Cell Malignancies
Brief Title: Rituximab in Treating Patients Undergoing Donor Peripheral Blood Stem Cell Transplant for Relapsed or Refractory B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Maloney, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2226.00; NCI-2010-00107 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2226; 2226.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P01CA078902 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: B-cell Adult Acute Lymphoblastic Leukemia; B-cell Childhood Acute Lymphoblastic Leukemia; B-cell Chronic Lymphocytic Leukemia; Childhood Burkitt Lymphoma; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Recurrence; Leukemia, Hairy Cell; Waldenstrom Macroglobulinemia | interventions — Rituximab; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (rituximab pre- and post-transplant) (Experimental): Patients receive rituximab IV, pre- and post-transplant, on days -3, 10, 24, and 38. Patients undergo donor peripheral blood stem cell transplant on day 0. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Procedure: peripheral blood stem cell transplantation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Procedure: peripheral blood stem cell transplantation — Undergo nonmyeloablative allogeneic peripheral blood/hematopoietic stem cell transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo nonmyeloablative allogeneic peripheral blood/hematopoietic stem cell transplantation
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies giving rituximab before and after a donor peripheral blood stem cell transplant in patients with B-cell lymphoma that does not respond to treatment (refractory) or has come back after a period of improvement (relapsed). Monoclonal antibodies, such as rituximab, can interfere with the ability of cancer cells to grow and spread. Giving rituximab before and after a donor peripheral blood stem cell transplant may help stop cancer from coming back and may help keep the patient's immune system from rejecting the donor's stem cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of addition of peri-transplant rituximab on relapse rate at 18 months after non-myeloablative allogeneic hematopoietic cell transplant (HCT) for cluster of differentiation (CD)20+ B-cell malignancies.

SECONDARY OBJECTIVES:

I. To determine overall and progression-free survival and non-relapse mortality.

II. To determine the incidence and severity of acute and chronic graft-versus-host disease (GVHD).

III. To determine the rate of graft rejection and graft failure.

IV. To determine the time to engraftment.

V. To determine the incidence of serious adverse events with the addition of rituximab.

VI. To evaluate the pharmacokinetics of rituximab in the setting of non-myeloablative allogeneic HCT.

VII. To describe donor and host polymorphisms of the FC gamma receptor IIIa (FCg RIIIA) and CD32 and evaluate their impact on disease response and relapse.

OUTLINE:

Patients receive rituximab intravenously (IV), pre- and post-transplant, on days -3, 10, 24, and 38. Patients undergo donor peripheral blood stem cell transplant on day 0. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 18 months and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* With a diagnosis of CD20-expressing B-cell malignancy of any histologic type or grade for whom non-myeloablative allogeneic transplant is considered an appropriate treatment option
* Who are enrolled on a non-myeloablative allogeneic HCT protocol employing total-body irradiation (TBI)-based conditioning of =< 4.5 Gy, with or without fludarabine; this protocol may be used as an adjunct to the allogeneic arm of a tandem autologous/allogeneic transplant protocol, provided the allogeneic conditioning meets the above criteria
* Receiving unmodified peripheral blood mononuclear cell graft products
* With an appropriate related or unrelated donor; human leukocyte antigen (HLA)-haploidentical donors are excluded
* Able to give informed consent (if >= 18 years of age), or with a legal guardian capable of giving consent (if < 18 years of age)

Exclusion Criteria:

* Ineligible for non-myeloablative allogeneic HCT
* Receiving an HLA-haploidentical allograft
* Who are fertile but unwilling to use contraception during and for at least 12 months after HCT
* Females who are pregnant or breast-feeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Shadman M, Maloney DG, Storer B, Sandmaier BM, Chauncey TR, Smedegaard Andersen N, Niederwieser D, Shizuru J, Bruno B, Pulsipher MA, Maziarz RT, Agura ED, Hari P, Langston AA, Maris MB, McSweeney PA, Storb R, Sorror ML. Rituximab-based allogeneic transplant for chronic lymphocytic leukemia with comparison to historical experience. Bone Marrow Transplant. 2020 Jan;55(1):172-181. doi: 10.1038/s41409-019-0660-8. Epub 2019 Sep 3. PMID 31481800

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Rituximab Pre- and Post-transplant)
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Rituximab Pre- and Post-transplant)
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 58
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 63

OUTCOME MEASURES:

1. Primary Outcome: Disease Relapse Rate
Description: Number of patients with relapsed/progressive disease post-transplant. The effectiveness of pre- and post-transplant rituximab in decreasing the rate of relapse will be evaluated.
Time Frame: At 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab Pre- and Post-transplant)
Number analyzed (Participants) | 63
Participants | 18

2. Secondary Outcome: Incidence and Severity of Acute and Chronic GVHD Evaluated Per an Adapted Version of Common Terminology Criteria for Adverse Events (CTCAE) Version 2.0
Description: Number of patients who developed acute/chronic GVHD post-transplant. A chronic GVHD diagnosis ≥1 manifestation that is distinctive for chronic GVHD, as opposed to acute GVHD.
  aGVHD Stages
  Skin:
  a maculopapular eruption involving < 25% BSA a maculopapular eruption involving 25 - 50% BSA generalized erythroderma generalized erythroderma with bullous formation and often with desquamation
  Liver:
  bilirubin 2.0 - 3.0 mg/100 mL bilirubin 3 - 5.9 mg/100 mL bilirubin 6 - 14.9 mg/100 mL bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: Through day +100 after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab Pre- and Post-transplant)
Number analyzed (Participants) | 63
Participants | 17

3. Secondary Outcome: Overall Survival and Progression-free Survival
Description: Number of patients surviving and number of patients surviving without progressive/relapsed disease, post-transplant.
Time Frame: At 6 months and then every year thereafter, up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab Pre- and Post-transplant)
Number analyzed (Participants) | 63
Participants
  PFS - 6 Months | 48
  PFS - 1 Year | 39
  PFS - 1.5 Years | 34
  OS - 6 Months | 52
  OS - 1 Year | 44
  OS - 1.5 Years | 36

4. Secondary Outcome: Rate of Graft Rejection and Graft Failure
Description: Number of patients experiencing graft rejection and/or graft failure
Time Frame: 18 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Rituximab Pre- and Post-transplant)
Number analyzed (Participants) | 63
Participants
  Graft Rejection | 1
  Graft Failure | 0

5. Secondary Outcome: Time to Engraftment
Description: Median time from transplant to engraftment.
Time Frame: 18 Months
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Rituximab Pre- and Post-transplant)
Number analyzed (Participants) | 63
Days | 10 [0 to 48]

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Arm/Group | Treatment (Rituximab Pre- and Post-transplant)
Serious Adverse Events (participants affected / at risk) | 5/63
Other Adverse Events (participants affected / at risk) | 15/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Rituximab Pre- and Post-transplant) (N=63)
Multiple Pulmonary Emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Suspected Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death Due to Infection (Infections and infestations) | 2 (2)
Sepsis and Tachycardia (Infections and infestations) | 1 (1)
Sepsis, Respiratory Failure, Mental Status Change (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Rituximab Pre- and Post-transplant) (N=63)
ARDS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Elevated Bilirubin (Hepatobiliary disorders) | 4 (4)
Elevated Creatinine (Renal and urinary disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes